CLINICAL TRIAL: NCT03738202
Title: Multifaceted Intervention Package for Protection Against Cotton Dust Exposure Among Textile Workers - a Cluster Randomised Controlled Trial
Brief Title: Multifaceted Intervention for Protection Against Cotton Dust Exposure Among Textile Workers
Acronym: MultiTex-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Wellcome Trust (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Asaad Ahmed Nafees, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MultiTex-RCT
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Occupational Diseases; Occupational Lung Disease
Keywords: Randomized controlled trial; Textile industry; Cotton fiber; Byssinosis
MeSH Terms: conditions — Occupational Diseases; Byssinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Multifaceted intervention package will be implemented at textile mills in the intervention arm.
  Interventions: Behavioral: Multifaceted intervention package
- Control (No Intervention): No intervention will be provided to mills in the control arm.

INTERVENTIONS:
Behavioral: Multifaceted intervention package — Multifaceted intervention package will comprise following strategies:
  1. Initial training for all workers and managers on occupational health and safety (OHS)
  2. Follow-up refresher sessions every three months
  3. Formation of workplace committees (including worker representatives) to draw up, agree and promote a health and safety plan that includes wet mopping, safe disposal of cotton dust, and the use of simple face masks, as well as further publicity about the risks from cotton dust.
  4. Provision of adequate supplies of face masks to support the health and safety plan
  Arms: Intervention

SUMMARY:
Textile workers are exposed to various harmful substances during work, including cotton dust, which is the dust present in air during the handling or processing of cotton. Previous research found a link between cotton dust exposure and impaired respiratory health. This study will comprise of administration and workers' training regarding preventive measures for protection against respiratory illnesses. Workers will be provided free, disposable face masks and measures to reduce cotton dust exposure will be introduced at the textile mills. The study would then determine the effectiveness of this intervention on reduction in cotton dust levels in the mills, and improvement in respiratory health of workers. This study would help the cotton textile workers and managers reduce the health hazards of cotton dust exposure and also guide researchers from Pakistan and other low-resource countries towards developing relevant strategies for health protection of these workers.

DETAILED DESCRIPTION:
The textile, clothing and footwear sector provides employment to more than 60 million people worldwide, mostly in developing countries. Pakistan's textile industry accounts for 8.5% of the national GDP and employs around 40% of the industrial workforce. High burden of respiratory illnesses, including byssinosis and lung function decrements has been reported among cotton textile workers in developing countries and previous work undertaken by Dr Nafees found a high burden in Pakistan. Dr Nafees recently implemented an interventional study designed to improve workers' knowledge, attitude and practices and respiratory health, and reduce dust exposure at cotton textile mills through a multifaceted intervention (MultiTex pilot study). The preliminary findings from the pilot were helpful in improving the overall design and implementation of a larger and more definitive study (cluster randomised controlled trial). The aim of the trial would be to determine the effectiveness of a multifaceted interventional package for improvement in reducing dust levels at the cotton textile mills as well as improvement in respiratory health of textile workers.This study will add important context-specific knowledge regarding preventive strategies in cotton mills with policy implications for Pakistan and other developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for textile mills:
* Mills from the formal sector will be included.
* Mills which have either spinning or weaving sections, or both.
* Mills that have at least 50-100 workers (primarily labourers/machine operators) in the spinning and weaving sections.
* Mills with a more stable working population will be preferred.
* Willingness of management to participate in planning and implementation of the study.
* Inclusion criteria for textile workers:
* Those ≥18 years and employed in the bale opening, blowing, carding, spinning, weaving and waste recycling sections (and related sub-sections).

Exclusion Criteria:

* Textile workers from the wet-processing areas as well as support or administrative staff will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2031 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Changes in cotton dust personal exposure levels expressed as mg/m3 | 24 months
  Will be assessed through the use of IOM samplers
Changes in the prevalence of respiratory symptoms | 24 months
  Will be assessed through MRC respiratory questionnaire; symptoms include chest tightness, cough, phlegm, chronic bronchitis, wheezing and shortness of breath.
Changes in Forced Expiratory Volume in first second (FEV1) measured in in ml | 24 months
  Will be assessed through spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Asaad A Nafees, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
This may be possible at the conclusion of the study and would depend on the guidelines of the funding agency and the publishing journal(s).

REFERENCES:
- [Background] Nafees AA, De Matteis S, Kadir MM, Burney P, Coggon D, Semple S, Cullinan P. MultiTex RCT - a multifaceted intervention package for protection against cotton dust exposure among textile workers - a cluster randomized controlled trial in Pakistan: study protocol. Trials. 2019 Dec 16;20(1):722. doi: 10.1186/s13063-019-3743-3. PMID 31842937
- [Background] Nafees AA, Matteis S, Burney P, Cullinan P. Contemporary Prevalence of Byssinosis in Low- and Middle-Income Countries: A Systematic Review. Asia Pac J Public Health. 2022 Jul;34(5):483-492. doi: 10.1177/10105395211073051. Epub 2022 Jan 24. PMID 35073782
- [Result] Nafees AA, Iqbal AR, Cullinan P, De Matteis S, Burney P, Semple S. Use of Low-Cost Particle Counters for Cotton Dust Exposure Assessment in Textile Mills in Low- and Middle-Income Countries. Ann Work Expo Health. 2022 Apr 22;66(4):537-542. doi: 10.1093/annweh/wxab102. PMID 34791042
- [Result] Nafees AA, Muneer MZ, De Matteis S, Amaral A, Burney P, Cullinan P. Impact of using different predictive equations on the prevalence of chronic byssinosis in textile workers in Pakistan. Occup Environ Med. 2022 Apr;79(4):242-244. doi: 10.1136/oemed-2021-107680. Epub 2021 Nov 19. PMID 34799440
- [Result] Nafees AA, Muneer MZ, Irfan M, Kadir MM, Semple S, De Matteis S, Burney P, Cullinan P. Byssinosis and lung health among cotton textile workers: baseline findings of the MultiTex trial in Karachi, Pakistan. Occup Environ Med. 2023 Mar;80(3):129-136. doi: 10.1136/oemed-2022-108533. Epub 2023 Jan 30. PMID 36717255